CLINICAL TRIAL: NCT04600037
Title: Effectiveness of Pregabalin Treatment for Trigger Points in Patients With Comorbid Myofascial Pain Syndrome and Fibromyalgia Syndrome: a Randomized Controlled Trial
Brief Title: Pregabalin Treatment for Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FSMEAH-KAEK 2014/20
Record Dates: First submitted 2020-10-18; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Myofascial Pain Syndrome
Keywords: fibromyalgia, trigger point, myofascial pain, pregabalin
MeSH Terms: conditions — Myofascial Pain Syndromes; Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients received pregabalin (target dose 300 mg/day) and exercise therapy (stretching exercises for the trapezius muscle). Patients were instructed to perform 10 repetitions three times a day., 3 months
  Interventions: Drug: Pregabalin 150mg
- Group 2 (No Intervention): Patients received exercise therapy alone (stretching exercises for the trapezius muscle). Patients were instructed to perform 10 repetitions three times a day., 3 months

INTERVENTIONS:
Drug: Pregabalin 150mg — Patients in group I received pregabalin at a dose of 75 mg twice daily during the first week that was increased to 150 mg twice daily thereafter and maintained at that level for 12 weeks.
  Patients in two groups received exercise therapy (stretching exercises for the trapezius muscle). Patients were instructed to perform 10 repetitions three times a day., 3 months
  Arms: Group 1

SUMMARY:
Myofascial pain syndrome (MPS) is a common problem in the general population. MPS should not be a local/peripheral painful syndrome and considered to be a syndrome of central sensitivity. We aimed to investigate the effect of pregabalin in patients with MPS in this study

DETAILED DESCRIPTION:
We randomized 40 patients into two groups, and 17 patients per group completed the study. Patients in group I received pregabalin and exercise therapy, whereas those in group II received exercise therapy alone. All patients were evaluated as follows: for pain by VAS; trigger-point pressure pain threshold-(PPT) by algometry; neuropathic pain using DN4 and quality of life with the SF36. Evaluations were performed pretreatment and at the end of the first and third months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed fibromyalgia syndrome,
* Patients who were also diagnosed as cervical myofascial pain syndrome based on the upper trapezius muscle

Exclusion Criteria:

* Patients who had received dry needling or local anesthetic injection to trigger point in the dominant upper trapezius muscle within 3 months of the start of the study.
* renal insufficiency,
* impaired liver function,
* malignancy,
* pregnancy
* infections,
* history of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04-26 (Actual); Primary Completion 2014-07-26 (Actual); Study Completion 2015-01-26 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 3 months
  VAS is psychometric measuring instrument designed to document the characteristics of disease-related symptom severity in each patient and use this to achieve a rapid classification of symptom severity and disease control. Patients were instructed to rate their pain between 0 and 10
Pressure pain thresholds (PPT) assessment | 3 months
  We assessed PPTs in upper trapezius trigger points with an algometer in all patients. PPT is defined as the minimal amount of pressure required to change a sensation of pressure to pain. An electronic algometer (Baseline Push Pull Force Gauge) was used, which consisted of a metal piston with a 1-cm circular rubber tip. Pressure measurements were recorded as kilograms per square centimeter (kg/cm2) with the patient in a seated position. The algometer was placed at a selected trigger point with the metal rod perpendicular to the surface of the skin, the pressure applied to the muscles was increased at a rate of approximately 1 kg per second, and the patient was instructed to state when pain was perceived. This procedure was repeated three times per patient, with 1-minute intervals. The mean of three trials (intra-examiner reliability) was calculated and used for the main analysis. If trigger points were in both upper trapezius muscle, the dominant side was evaluated.
DN4 - Questionnaire (DN4) | 3 months
  DN4 was used to evaluate neuropathic pain. DN4 is used to identify neuropathic pain and consists of ten questions. Seven questions are concerned with symptoms and three are concerned with clinical findings. Symptoms assessed are burning, painful cold, electric shocks, tingling, pins and needles, numbness, and itching. The physician assesses whether there is reduced sensation (hypoesthesia) to touch or pinprick, and if light brushing increases or causes pain (allodynia) by examination. Each item is scored "yes" (1 point) or "no" (0 points). If the total score is ≥4, the pain is likely to be neuropathic
Short Form-36 (SF36) | 3 months
  The SF36 is a self-reported questionnaire widely used to measure quality of life. The questions are summarized into eight scales: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems, and mental health. The initial four items form the physical component summary measuring physical health domains, while the latter four items form the mental component summary measuring mental health domains. Scores can range from 0 (worst health status) to 100 (best health status) per domain. Higher scores indicate better health status for the calculated sub item

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Silte Karamanlioglu, MD, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital; Duygu Geler Kulcu, prof, Study Director — Haydarpaşa Numune Training and Research Hospital; Gulcan Ozturk, MD, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Pinar Akpinar, Assoc prof, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Feyza Unlu Ozkan, Assoc prof, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Ilknur Aktas, Prof, Study Chair — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karamanlioglu DS, Geler Kulcu D, Ozturk G, Akpinar P, Unlu Ozkan F, Aktas I. Effectiveness of pregabalin treatment for trigger points in patients with comorbid myofascial pain syndrome and fibromyalgia syndrome: a randomized controlled trial. Somatosens Mot Res. 2021 Dec;38(4):327-332. doi: 10.1080/08990220.2021.1977265. Epub 2021 Sep 20. PMID 34544324